CLINICAL TRIAL: NCT01909856
Title: The Efficacy and Safety of Palonosetron in Preventing the Gastrointestinal Reactions Induced by 3-day Highly Emetogenic Chemotherapy
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Jiangsu Simcere Pharmaceutical Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Prevention
Other Study IDs: sim-palonosetron
Record Dates: First submitted 2013-07-22; First posted 2013-07-29 (Estimated); Last update posted 2015-12-04 (Estimated); Status verified 2015-11

CONDITIONS: Cancer
MeSH Terms: conditions — Neoplasms | interventions — Palonosetron; Granisetron; Dexamethasone; Cisplatin

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Arm1 (Experimental): 1st cycle Palonosetron, 2nd cycle Granisetron
  Interventions: Drug: Palonosetron; Drug: Granisetron; Drug: Dexamethasone; Drug: Cisplatin
- Arm2 (Experimental): 1st cycle Granisetron, 2nd cycle Palonosetron
  Interventions: Drug: Palonosetron; Drug: Granisetron; Drug: Dexamethasone; Drug: Cisplatin

INTERVENTIONS:
Drug: Palonosetron — Palonosetron 0.25mg d1,d3
Drug: Granisetron — Granisetron 3mg d1-3
Drug: Dexamethasone — Dexamethasone 10mg d1-3
Drug: Cisplatin — 3-day chemotherapy regimens including cisplatin, cisplatin: 25mg/m2 d1-3

SUMMARY:
This study is to assess the efficacy and safety of palonosetron in preventing the acute and delayed emesis induced by 3-day highly emetogenic chemotherapy. A double-blind, crossover design is used and granisetron is the positive control.

ELIGIBILITY:
Inclusion Criteria:

* Patients diagnosed with malignant tumors who can receive 3-day chemotherapy regimens defined by the protocol;
* The two-cycle sequential chemotherapy must be the same in drugs, dosage, sequence and routes of administration;
* Patients are prohibited from any other chemotherapy drugs during the study, as well as other antiemesis, sedative and psychotropic drugs within 5 days after chemotherapy;
* Life expectancy ≥ 3 months;
* Adequate hematologic function;
* Adequate hepatic function;
* Adequate renal function;
* At least 2 weeks away from the last chemotherapy;
* Patients signed written informed consent.

Exclusion Criteria:

* Pregnant or lactating women;
* History of anticipatory vomiting;
* Radiation therapy on the abdomen or pelvis within one week prior to study entry;
* Concomitant use of other drugs which may affect the antiemetic effects (such as omeprazole, amifostine, etc.);
* Patients with gastrointestinal obstruction;
* Patients with severe heart disease, liver or renal disease, or metabolism disorders;
* Patients with epilepsy or using sedative or psychotropic drugs;
* Patients with diabetes or with contraindication for corticosteroids;
* Patients who received antiemetic drugs or experienced nausea or vomiting within 24 hours prior to study entry;
* Patients with brain metastasis or intracranial hypertension;
* Hypersensitivity to 5-HT3 receptor antagonist;
* Patients with active infection;
* Other conditions that the investigator considered as unsuitable for chemotherapy;
* Subjects participating in other clinical trials.

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 92 (Actual)
Dates: Start 2011-10; Primary Completion 2014-04 (Actual); Study Completion 2014-06 (Actual)

PRIMARY OUTCOMES:
Complete Response(CR) within 24-120 hours after chemotherapy | 24-120 hours

SECONDARY OUTCOMES:
CR within 0-120 hours after chemotherapy | 0-120 hours
CR within 0-24 hours after chemotherapy | 0-24 hours
Incidence of Adverse events | up to 3 months

CONTACTS AND LOCATIONS:
Overall Officials: Shiying Yu, MD, Principal Investigator — Tongji Hospital
Locations (1):
- Tongji Hospital,Tongji Medical College, Huazhong University of Science and Technology, Wuhan, Hubei, China